CLINICAL TRIAL: NCT00098241
Title: Multicenter Trial of the Safety & Efficacy of Certican in Pediatric de Novo Renal Transplant Patients
Brief Title: Safety & Efficacy of Certican in Pediatric de Novo Renal Transplant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001AB351; RAD/Certican
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplantation
Keywords: pediatric; renal; transplant recipients; de novo; De novo renal pediatric transplant
MeSH Terms: interventions — Everolimus

INTERVENTIONS:
Drug: Certican

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of RAD001 (Certican) administered to pediatric renal transplant recipients, and to provide additional safety data.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients no more than 16 years of age.
* Patients receiving a primary cadaveric or non-HLA identical living donor (related or unrelated) renal transplant.
* The graft must be functional within 48 hours post transplantation.

Exclusion Criteria:

* Cold ischemia time greater than 40 hours.
* Patients who are recipients of multiple solid organ transplants, including dual and en bloc kidneys, or who have previously received transplanted organs.
* Patients with panel reactive T cell antibodies of 50 % or higher at the last assessment before transplantation.

Ages: 1 Week to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2000-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability at 6 and 12 Months as measured by adverse events, laboratory abnormalities and infections.

SECONDARY OUTCOMES:
Efficacy at 6 and 12 Months as measured by rejection, graft loss, death and loss to follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (2):
- Columbus Children's Hospital, Columbus, Ohio, United States
- Dienst Pediatrie UZ Gasthuisberg, Herestraat 49, Leuven, Belgium

REFERENCES:
- [Result] Ettenger RB, Grimm EM. Safety and efficacy of TOR inhibitors in pediatric renal transplant recipients. Am J Kidney Dis. 2001 Oct;38(4 Suppl 2):S22-8. doi: 10.1053/ajkd.2001.27838. PMID 11583941